CLINICAL TRIAL: NCT01856985
Title: The Acceptability of an Out-patient Regimen of Medical Abortion With Mifepristone and 800 Mcg Misoprostol Administered Buccally or Sublingually at 78-84 Days Gestation: Two Pilot Studies
Brief Title: Acceptability of an Out-patient Regimen of Medical Abortion With Mifepristone and 800 Mcg Misoprostol Administered at 78-84 Days Gestation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1010
Record Dates: First submitted 2013-04-30; First posted 2013-05-20 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Medical Abortion
Keywords: Medical abortion; Misoprostol; Mifepristone
MeSH Terms: interventions — Misoprostol; Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Misoprostol at clinic (Experimental): Eligible women will receive 200 mg mifepristone to be administered at home or at the clinic and will receive either 800 µg misoprostol buccally (study 1) or 800 µg misoprostol sublingually (study 2) to self administer at home.
  Participants will be asked to return to the hospital 14 days later for a follow-up visit.
  Interventions: Drug: Misoprostol; Drug: Mifepristone

INTERVENTIONS:
Drug: Misoprostol
Drug: Mifepristone

SUMMARY:
These pilot studies are designed as open label studies to investigate the acceptability of 200 mg mifepristone followed 24-48 hours later by either 1) 800 µg misoprostol administered buccally or 2) 800 µg misoprostol administered sublingually for medical abortion in gestations 78-84 days' LMP. They will be done consecutively.

Findings from the pilot studies will guide the development of a larger, multi-site study to investigate the efficacy of outpatient medical abortion regimens for women with gestations from 78 - 84 days LMP. In that end, the pilots seek to collect information on the acceptability of an outpatient medical abortion regimen of 200 mg oral mifepristone followed by either 800 mcg misoprostol delivered either buccally or sublingually safe acceptable? Women's rating of the tolerability of any side effects will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Seeking abortion services
* Have an intrauterine pregnancy 78 days through 84 days' LMP
* Be willing and able to sign consent forms
* Agree to comply with study procedures and visit schedule
* Be living with 30 minutes from the hospital

Exclusion Criteria:

* Does not meet the inclusion criteria outlined above

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percentage of women who have undergone a successful abortion | 2 weeks

SECONDARY OUTCOMES:
Women's acceptability of the assigned method. | 2 weeks
Side effects | 48 hours
  Side effects include nausea, vomiting, pain, diarrhea, fever. Asked women to rank as none, mild, moderate, severe. Used an acceptability scale (Very Acceptable v. Acceptable v. Neutral v. Unacceptable v. Very unacceptable v. Don't know) to ascertain acceptability among women

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Jennifer Blum, MPH, Principal Investigator — Gynuity Health Projects; Nguyen Thu Nhu Ngoc, MD, Principal Investigator — Center for Research and Consultancy in Reproductive Health; Dina F Abbas, Principal Investigator — Gynuity Health Projects
Locations (1):
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam